CLINICAL TRIAL: NCT02764684
Title: The Effect of Probiotics on Microbial Translocation and Inflammation in HIV-infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Susanne Dam Nielsen, MD, Associate Professor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 43771
Record Dates: First submitted 2015-11-04; First posted 2016-05-06 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: HIV
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIV-infected patients (Experimental): Probiotics (lactobacillus rhamnosus)
  Interventions: Drug: Probiotic

INTERVENTIONS:
Drug: Probiotic — The probiotic strain Lactobacillus rhamnosus will be self-administrated twice a day, one capsule in the morning and one in the evening for eight weeks.
  Other Names: Lactobacillus rhamnosus

SUMMARY:
Objective:

In this study the investigators aim at investigating:

1. probiotics ability to modulate the microbiome and microbial translocation,
2. if probiotics affect the level of cholesterol, triglycerides as markers of cardiovascular risk factors and
3. if a reduction of microbial translocation is associated with a reduction of inflammation in the gastro-intestinal tract.

Design:

The study is a prospective clinical intervention trial of 40 HIV-infected patients.

Method:

The investigator will administer the bacteria Lactobacillus Rhamnosus in capsular form to each patient 2 times a day in 8 weeks. At baseline and at the 8th week of the intervention, the investigators will collect blood samples, feces samples and make a positron emission tomography-magnetic resonance scans.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* confirmed HIV
* no HIV treatment
* cluster of differentiation 4+ cell count over 350

Exclusion Criteria:

* antibiotic or probiotic in last 2 month
* drugs that influence gut motility
* diabetes
* Inflammatory bowel disease
* cancer
* autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
change in Lipopolysaccharide (unit= endotoxin unit/mL) from baseline after intervention | Will be measured before and after eight weeks of intervention.
  will be measured in plasma samples

SECONDARY OUTCOMES:
change in soluble cluster of differentiation 14 (unit (ng/mL) from baseline and eight weeks after intervention. | Will be measured before and after eight weeks of intervention.
  will be measured in plasma samples
change in inflammation around the gut measured with positron emission tomography-magnetic resonance scans of the abdomen ( size of the lymph nodes and positron emission tomography-activity) | Will be measured before and after eight weeks of intervention.
  positron emission tomography-magnetic resonance scans of the abdomen before an after intervention
Changes in of high sensitive C-reactive protein (unit mg/l) from baseline and after eight weeks of intervention | Will be measured before and after eight weeks of intervention.
  will be measured in plasma samples
Changes in measures of cytokines unit (pg/ml) at baseline and after eight weeks of intervention | Will be measured before and after eight weeks of intervention.
  will be measured in plasma samples
Changes in the gut microbiota composition (454 pyrosequencing of fecal samples) from baseline to eight weeks after intervention (end of study) | Will be measured before and after eight weeks of intervention.
  stool-samples will be collected an analyzed by deep sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Susanne D Nielsen, MD, DMSc, Principal Investigator — Rigshospitalet, danmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The investigator plan to publish data in an article when the study is completed